CLINICAL TRIAL: NCT00613873
Title: A Model Program for Increasing Use of Screening Colonoscopy Among Minority Women and Men
Brief Title: Use of Screening Colonoscopy Among Minority Women and Men
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: North General Hospital, New York (Other); Ralph Lauren Center for Cancer Care and Prevention (Other)
Responsible Party: Moshe Shike, M.D., Memorial Sloan Kettering Cancer Center
Other Study IDs: 03-066
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Colorectal Screening
Keywords: colonoscopy
MeSH Terms: interventions — Colonoscopy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Women participating in a community based mammography or cervical screening program will also participate in colonoscopy screening. Participation will be measured by stating an interest in colorectal cancer screening and then following through with colonoscopy screening. Furthermore we will assess whether those complying with colonoscopy will also recommend colonoscopy screening for their spouses or household members.
  Interventions: Procedure: Colonoscopy and Questionnaire

INTERVENTIONS:
Procedure: Colonoscopy and Questionnaire — Pt is asked to complete attitude and belief questionnaire then have a Colonoscopy. Then within 6 weeks post colonoscopy a final telephone interview.

SUMMARY:
Colorectal cancer is a cancer in the colon or rectum. Routine screening can find it at an early stage, when it has a much higher chance of cure. Screening can also help to find polyps. These are mushroom shaped growths that could turn into cancer. A polyp can be removed before it turns into cancer. Even though screening can save lives, not enough people in the country are having it. This is especially true in Harlem. Harlem has a higher rate of deaths from this cancer than other places in the U.S. because too many people do not get screened. By the time a person has symptoms, the cancer may be at a late stage, when it is much harder to cure.

We are doing this study to see if we can increase the number of people in Harlem who get screened. We plan to tell women about the screening when they have a mammogram or pap test. We will also ask them what they know and think about colorectal cancer. And, we will see if they get other members of their household to be screened.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 50
* Availability by telephone

Exclusion Criteria:

* History of colorectal cancer screening (fecal occult blood testing annually for last 3 years; colonoscopy within the last 10 years)
* History of colorectal cancer
* Serious illness which precludes colonoscopy (severe heart disease; severe pulmonary disease; uncontrolled diabetes; uncontrolled hypertension; other medical contraindication)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigators or research team at Memorial Sloan-Kettering Cancer Center(MSKCC). The study will be offered to all eligible women who come for breast or cervical cancer screening at The Breast Examination Center of Harlem during the study period
Sampling Method: Non-Probability Sample
Enrollment: 611 (Actual)
Dates: Start 2003-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of using a community screening mammography center to recruit minority women form a low income community to undergo colorectal cancer screening (CRCS). | conclusion of the study

SECONDARY OUTCOMES:
Identify individual level barriers (demographic, financial, and psychological) to CRCS among minority women who are already participating in screening for another cancer (breast or cervical) | conclusion of the study
Determine the feasibility of promoting CRCS among spouses (and other members of the household) of minority women who have undergone screening colonoscopy. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Shike, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Breast Examination Center of Harlem, New York, New York

REFERENCES:
- [Derived] Shike M, Schattner M, Genao A, Grant W, Burke M, Zauber A, Russo L, Cuyjet V. Expanding colorectal cancer screening among minority women. Cancer. 2011 Jan 1;117(1):70-6. doi: 10.1002/cncr.25566. Epub 2010 Oct 25. PMID 21170901
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org